CLINICAL TRIAL: NCT06049784
Title: Prelabor Maternal Pushing Training Using Visual Biofeedback by a Self-operated Ultrasound Device
Brief Title: Prelabor Visual Biofeedback by a Self-operated Ultrasound Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Sharon Perlman, Senior attending physician, Proffesor of Obstetrics and Gynecology, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RMC-0400-21
Record Dates: First submitted 2023-09-01; First posted 2023-09-22 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Obstetric Labor Complications; Obstetric Trauma
Keywords: Visual Biofeedback; Self Operated Ultrasound device; Second stage of labor; Trans Perineal Ultrasound
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Intervention Model Description: Parallel assignment Randomised Control Trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will collect the data from the files without knowing the participants' group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Visual Biofeedback using self operated home ultrasound device (Experimental): Sonographic fetal weight and biophysical profiles will be done at the hospital clinic. A single ultrasound biofeedback session using trans-perineal Ultrasound (TPU) will guide maternal pushing. The process includes (a) Ultrasound assessing fetal head descent with the screen facing the provider, measuring the angle of progression (AOP); (b) Explaining anatomical landmarks to the patient; (c) Repeat AOP measurement with the screen facing the patient for biofeedback; (d) Reassess with the screen turned away.
  Participants will receive a handheld home ultrasound device, learning to perform self-biofeedback at home, ideally twice a week, up to 4 times. Session records will be sent electronically to the sonographer for assessment and feedback.
  All groups will complete questionnaires three times: (1) baseline, (2) about two weeks later (after home biofeedback training), and (3) six to eight weeks postpartum.
  Interventions: Device: Visual Biofeedback using self operated home ultrasound device
- Visual biofeedback at the Hospital (Active Comparator): A sonographic fetal weight estimate and biophysical profile will occur at the hospital clinic for all patients. A single ultrasound-based biofeedback session will employ TPU for maternal pushing guidance. This process involves (a) Assessing fetal head descent with ultrasound to measure the angle of progression (AOP) during rest and pushing; (b) Explaining anatomical landmarks to the patient; (c) Repeating the AOP measurement as biofeedback; (d) Reassessing with the screen turned away.
  Participants will complete questionnaires three times: (1) baseline, (2) two weeks later, and (3) six to eight weeks postpartum.
  Interventions: Device: Visual Biofeedback using ultrasound at hospital
- Control / Standard care - Obstetrical ultrasound only (No Intervention): A sonographic estimated fetal weight and biophysical profile will be performed in the hospital.
  The participant will fill in questionnaires at three time points: (1) at baseline, before the ultrasound examination; (2) about two weeks later (i.e., after completing the self-operated visual biofeedback training at home, or at an equivalent time for the other two groups); (3) six to eight weeks postpartum.

INTERVENTIONS:
Device: Visual Biofeedback using self operated home ultrasound device — participants will receive a handheld home ultrasound device, learning to perform self-biofeedback at home. Session records will be sent electronically to the sonographer for assessment and feedback.
  Arms: Visual Biofeedback using self operated home ultrasound device
Device: Visual Biofeedback using ultrasound at hospital — A single ultrasound biofeedback session using Transperineal Ultrasound will guide maternal pushing.
  Arms: Visual biofeedback at the Hospital

SUMMARY:
A substantial number of women report fear of childbirth and negative birth experiences. The objective of the study is to assess the efficacy of visual biofeedback before labor using a self-operated home ultrasound for maternal pushing training, which is expected to reduce fear of childbirth, increase perceived control during birth, prevent prolonged labor and the ensuing maternal and neonatal negative adverse outcomes, and prevent maternal post-traumatic stress symptoms. Intrapartum visual biofeedback provided by obstetricians during the second stage of labor has been shown to increase pushing efficiency and improve maternal obstetric and psychological outcomes. Previously, visual biofeedback has been implemented only in an in-hospital setting and, with one known exception, only during labor. A Mobile Self-Operated Home Ultrasound System has been reported as a feasible and reliable tool for obstetrical ultrasound. A randomized controlled trial will be conducted with three study groups of pregnant women (37-39 weeks of gestation): (1) Obstetrical ultrasound+visual biofeedback in-hospital and at home using self-operated ultrasound; (2) Obstetrical ultrasound+visual biofeedback in-hospital; (3) Obstetrical ultrasound only. Visual biofeedback by ultrasound will be performed by transperineal ultrasound, enabling the future mother to visualize the descent of the fetal head within the birth canal in response to her pushing effort. Follow-up will be conducted two weeks later and at six weeks postpartum. Positive results following the application of biofeedback by self-operated home ultrasound may change the paradigm for pre-labour sonographic education. Self-operated home ultrasound will also enable more comprehensive pre-labor ultrasound-based education and hopefully reduce adverse physical and psychological outcomes following childbirth.

DETAILED DESCRIPTION:
The primary goal of this study is to evaluate the effectiveness of visual biofeedback prior to labor, which involves a single session in the hospital combined with a self-administered home ultrasound to train mothers on pushing techniques during the second stage of labor. The approach integrates a one-time pre-labor training session at the clinic, as previously explored by Youssef et al. (2021), with a continued two-week intervention carried out by the participants at home. This method is anticipated to enhance the benefits noted in prior research. The study will examine the impact of this training intervention and then collect comprehensive data on both obstetric and psychological outcomes, which will include medical records and self-report questionnaires completed by the participants before and after childbirth. The intervention seeks to mitigate maternal and neonatal obstetric complications and other adverse outcomes. The specific objectives of this study are:

1. to decrease the duration of the second stage of labor, minimize medical interventions during labor, and lessen birth-related complications;
2. to alleviate prenatal fear of childbirth and bolster confidence in the birthing process;
3. to enhance perceived personal control during labor and increase satisfaction with the birthing experience;
4. to improve maternal-infant bonding and reduce incidences of post-traumatic stress symptoms;
5. to explore participants' experiences with the at-home, self-managed intervention and its effectiveness through semi-structured, in-depth interviews with a subset of the participants involved in this study.

ELIGIBILITY:
Inclusion Criteria:

* Nuliparity
* Singleton pregnancy
* Planned for vaginal delivery
* Low risk pregnancy
* Ability to fulfill a questionnaire

Exclusion Criteria:

* Multifetal gestation
* Contraindications for vaginal delivery (Placenta previa, Breech presentation etc.)
* High risk pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2023-12-31 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The length of the second stage of labour | up to 1 week after labor
  measure by time

SECONDARY OUTCOMES:
Mode of delivery | up to 1 week after labor
  Number of participants with spontaneous vaginal delivery or operative delivery (operative assisted - vacuum assisted/forceps, cesarean delivery)
OASIS - obstetrical anal sphincter injuries | up to 1 week after labor
  Number of Participants with severe perineal tear
Low neonatal APGAR score | up to 1 week after labor
  number of participants who delivered a neonate with APGAR score < 7 at 5 minutes after birth
NICU (neonatal intensive care unit) hospitalization | up to 1 week after labor
  number of participants who delivered a neonate transferred to the NICU
Fear of childbirth | up to 4 weeks before labor
  Number of participants who demonstrated fear of childbirth according to questionnaires
PTSS (post traumatic stress symptoms) | up to 3 months post partum
  Number of participants who demonstrated PTSS according to questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Perlman, MD, Principal Investigator — Rabin Medical Center, affiliated to the Tel Aviv University, Tel Aviv, Israel; Natav Hendin, MD, Principal Investigator — Rabin Medical Center, affiliated to the Tel Aviv University, Tel Aviv, Israel
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No
All collected data will be securely stored and used solely for research, analysis, and reporting within the scope of this study. Any results or findings that we may share with the scientific community or the public will be presented in aggregated, de-identified, and anonymized formats to protect participant privacy.
  Our primary focus is to use the gathered data for research purposes, and we do not anticipate sharing individual participant data beyond the confines of this study's objectives.

REFERENCES:
- [Background] Gilboa Y, Frenkel TI, Schlesinger Y, Rousseau S, Hamiel D, Achiron R, Perlman S. Visual biofeedback using transperineal ultrasound in second stage of labor. Ultrasound Obstet Gynecol. 2018 Jul;52(1):91-96. doi: 10.1002/uog.18962. Epub 2018 May 29. PMID 29155474
- [Background] Bellussi F, Alcamisi L, Guizzardi G, Parma D, Pilu G. Traditionally vs sonographically coached pushing in second stage of labor: a pilot randomized controlled trial. Ultrasound Obstet Gynecol. 2018 Jul;52(1):87-90. doi: 10.1002/uog.19044. Epub 2018 May 30. PMID 29532533
- [Background] Hadar E, Wolff L, Tenenbaum-Gavish K, Eisner M, Shmueli A, Barbash-Hazan S, Bergel R, Shmuel E, Houri O, Dollinger S, Brzezinski-Sinai NA, Sukenik S, Pardo A, Navon I, Wilk Y, Zafrir-Danieli H, Wiznitzer A. Mobile Self-Operated Home Ultrasound System for Remote Fetal Assessment During Pregnancy. Telemed J E Health. 2022 Jan;28(1):93-101. doi: 10.1089/tmj.2020.0541. Epub 2021 Mar 15. PMID 33729014
- [Background] Schlesinger Y, Hamiel D, Rousseau S, Perlman S, Gilboa Y, Achiron R, Frenkel TI. Preventing risk for posttraumatic stress following childbirth: Visual biofeedback during childbirth increases maternal connectedness to her newborn thereby preventing risk for posttraumatic stress following childbirth. Psychol Trauma. 2022 Sep;14(6):1057-1065. doi: 10.1037/tra0000558. Epub 2020 Feb 27. PMID 32105133